CLINICAL TRIAL: NCT06052241
Title: Artificial Intelligence-based Prescription of Personalized Scalp Cosmetics: Efficacy Results
Brief Title: Artificial Intelligence-based Prescription of Personalized Scalp Cosmetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B-2107-697-301
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Dandruff; Folliculitis
MeSH Terms: conditions — Dandruff; Folliculitis

STUDY DESIGN:
Intervention Model Description: prospective, single-center, pre-post comparative study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-treatment (Active Comparator): After treatment using shampoo and scalp serum personalized according to their Scalp Photographic Index Artificial Intelligence (SPI-AI)-defined scalp types
  Interventions: Drug: shampoos and scalp serums
- Pre-treatment (No Intervention)

INTERVENTIONS:
Drug: shampoos and scalp serums — shampoos and scalp serums personalized according to their SPI-AI-defined scalp types
  Arms: Post-treatment

SUMMARY:
The investigators aimed to evaluate whether they can be improved by an AI-based personalized prescription of scalp cosmetics.

ELIGIBILITY:
Inclusion Criteria:

1. healthy adults aged >19 years
2. presence of scalp-related discomfort (such as itching, a sensation of heat, dandruff, excessive sebum, dryness, pain, or pimple)

Exclusion Criteria:

1. presence of active infectious scalp diseases
2. history of treatment with topical or systemic steroids, oral immunosuppressants, topical or systemic antibiotics, or antifungal agents that could affect the scalp conditions, within 4 weeks prior to the baseline
3. difficulty understanding or following the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Total Scalp Photographic Index (SPI) score | week 4
  Change from the baseline in the total SPI score. The total SPI score (0-75 points) is the sum of the SPI score of five areas: vertex, anterior, posterior, right, and left. Higher SPI scores mean a worse condition, and larger changes from baseline in the total SPI score mean a better outcome.

SECONDARY OUTCOMES:
Total Scalp Photographic Index (SPI) score | week 8
  Change from the baseline in the total SPI score. The total SPI score (0-75 points) is the sum of the SPI score of five areas: vertex, anterior, posterior, right, and left. Higher SPI scores mean a worse condition, and larger changes from baseline in the total SPI score mean a better outcome.
Total Scalp Photographic Index (SPI) score | week 12
  Change from the baseline in the total SPI score. The total SPI score (0-75 points) is the sum of the SPI score of five areas: vertex, anterior, posterior, right, and left. Higher SPI scores mean a worse condition, and larger changes from baseline in the total SPI score mean a better outcome.
subjective improvement in scalp conditions | week 4
  proportion of participants achieving improvement in more than one item on the questionnaire
participant's satisfaction | week 4
  proportion of participants satisfied with the products

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Im Na, M.D, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: No